CLINICAL TRIAL: NCT04593069
Title: Long-term Cognitive Impairment in ICU Patients, Admitted for COVID-19 Pneumonia: a Single Centre, Prospective Cohort Study
Brief Title: The COGCOV Study in ICU Patients
Acronym: COGCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Dieter Mesotten, MD, Ziekenhuis Oost-Limburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: COGCOV
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Covid19; Cognitive Impairment
MeSH Terms: conditions — COVID-19; Cognitive Dysfunction | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Intervention Model Description: All patients enrolled in the study will be contacted to answer additional questions regarding cognitive impairment
Masking Description: masking is not applicable for this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COVID-19 patients (Other): Neurocognitive impairment in COVID-19 patients
  Interventions: Behavioral: Neurocognitive assessment

INTERVENTIONS:
Behavioral: Neurocognitive assessment — 6 months after admission to the intensive care unit of Ziekenhuis Oost-Limburg, the patients will be tested on cognitive impairment

SUMMARY:
Acute Respiratory Distress syndrome (ARDS) is a pulmonary systematic inflammatory response, leading to acute respiratory failure with hypoxia and/or hypercarbia. COVID-19 evokes a viral pneumonia, which may result in ARDS as well. It is not yet clear if COVID-19 disease behaves like the typical ARDS. Corona virus causes primarily deep hypoxia. Hypoxia, on its own, can lead to long term cognitive impairment. However, critical illness also affects long-term neurocognitive functioning. The investigators will be researching the possibility of long-term cognitive impairment in COVID-19 ICU patients, in comparison with reference values of a healthy population as well as the values measured in critically ill patients, admitted not only for respiratory reasons.

DETAILED DESCRIPTION:
The investigators will conduct a single centre, prospective cohort study. COVID-19 patients from the Ziekenhuis Oost-Limburg cohort will be contacted by phone 6 months after admission at the ICU. Patients will be asked to participate in a study surrounding long term symptoms of COVID-19. When consent is given by the patiënt, the experimenter will conduct a short questionnaire over the phone with the patient or relative that is present at the time of the call. If the participant is fluent in Dutch, the experimenter will ask permission to visit their home to conduct more testing.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the intensive care unit of Ziekenhuis Oost-Limburg
* Being hospitalized between March 2020 and May 2020, and therefore being admitted 6 months prior to the study
* The reason of hospitalization was COVID-19 disease

Exclusion Criteria:

* No willingness to participate, and therefore not having signed the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Neurocognitive impairment measured by RBANS | 6 months after admission at the intensive care unit
  the Repeatable Battery for the Assessment of Neuropsychological Statusis (RBANS) is a neuropsychological test that provides information about 5 domains of cognition (1) immediate and (2) delayed memory, (3) attention, (4) visuospatial construction and (5) language) and provides a total score. It is a test that takes about 30 minutes and consists of twelve tests. These are: (1) List Learning, (2) Story Memory, (3) Figure Copy, (4) Line Orientation, (5) Picture Naming, (6) Semantic Fluency, (7) Digit Span, (8) Coding, (9) List Recall, (10) List Recognition, (11) Story Recall and (12) Figure Recall. According to the RBANS manual, the possible values for the RBANS scores at the item, domain, and scale level are 0 to 89, 40 to 154, and 40 to 160

SECONDARY OUTCOMES:
Neurocognitive impairment measured by TMT | 6 months after admission at the intensive care unit
  Trail Making Test (TMT) is a test of executive functioning, visual search speed, scanning, speed of processing and mental flexibility. The total score is the time in seconds spent to complete each part.
Neurocognitive impairment by the short IQCODE | 6 months after admission at the intensive care unit
  The short IQCODE is a 16 question long questionnaire that assesses cognitive impairment in elderly patients. An informant is required to rate a patient's cognitive changes over a 10 year time period. Each question is scored from 1 (much improved over time) to 5 (much worse).

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Mesotten, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium